CLINICAL TRIAL: NCT04676750
Title: Mindfulness-baseret Forebyggelse og Sundhedsfremme i Den Sidste Del af Arbejdslivet
Brief Title: MBSR for Work Active Seniors
Acronym: MBSR6065
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 10
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Health Promotion and Stress Prevention
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Experimental): receives 8-week MBSR course
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- control (No Intervention): receives intervention after experiment finishes

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — yoga, meditation and psycho education
  Arms: MBSR

SUMMARY:
Testing Mindfulness-based Stress Reduction (MBSR) in 60-65 year old senior employees.

DETAILED DESCRIPTION:
Outcome measures: HRV, blood pressure, weight, structural and functional brain scans, questionnaire

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* psychosis

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
self-perceived stress | 2 years
  questionnaire

SECONDARY OUTCOMES:
Heart rate variability | 2 years
blood pressure | 2 years
weight | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dansk Center for Mindfulness, Aarhus, Brabrand, Denmark

IPD SHARING:
Plan to Share IPD: No